CLINICAL TRIAL: NCT04607668
Title: PRESERVE 1: A Phase 3 Randomized, Double-blind Trial of Trilaciclib Versus Placebo in Patients Receiving FOLFOXIRI/Bevacizumab for Metastatic Colorectal Cancer
Brief Title: Trilaciclib, a CDK 4/6 Inhibitor, in Patients Receiving FOLFOXIRI/Bevacizumab for Metastatic Colorectal Cancer (mCRC):
Acronym: PRESERVE1
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The Sponsor made the decision to terminate the study and complete the final analysis for available data.
Sponsor: G1 Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: G1T28-207
Record Dates: First submitted 2020-10-20; First posted 2020-10-29 (Actual); Results first posted 2024-11-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-10

CONDITIONS: Colorectal Cancer Metastatic; Myelosuppression-Adult; Chemotherapeutic Toxicity
Keywords: Colorectal Cancer; mCRC; colon; chemotherapy-induced myelosuppression; chemotherapy-induced neutropenia; chemotherapy-induced anemia; CDK 4/6 inhibitor; trilaciclib; FOLFOXIRI; bevacizumab; myelosuppression; cyclin-dependent kinase 4/6 inhibitor; myelopreservation; rectum; Preserve; PRESERVE 1
MeSH Terms: conditions — Colorectal Neoplasms | interventions — trilaciclib

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-Blinded Trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- trilaciclib + FOLFOXIRI/bevacizumab (Experimental): During Induction the following study drugs are administered on Day 1:
  Irinotecan - IV, Oxaliplatin - IV, Leucovorin- IV, Fluorouracil - continuous infusion (CI) over 46 to 48 hours beginning on Day 1, Bevacizumab - IV
  Following completion of Induction, patients will continue in Maintenance, where they will continue to receive trilaciclib per randomization allocation at study entry. Trilaciclib will be administered prior to infusional- 5FU/leucovorin/bevacizumab at the same dose and schedule used during Induction.
  Interventions: Drug: Trilaciclib
- placebo + FOLFOXIRI/bevacizumab (Placebo Comparator): The subjects in the placebo arm will follow the same schedule as the trilaciclib arm, but will receive placebo instead of trilaciclib.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Trilaciclib — Trilaciclib diluted in dextrose 5% in water or normal saline (sodium chloride solution 0.9%) administered by IV infusion over approximately 30 (±10) minutes no more than 4 hours prior to each Day 1 chemotherapy administration. Second dose of trilaciclib was administered on Day 2.
  Other Names: G1T28; CDK 4/6 inhibitor
  Arms: trilaciclib + FOLFOXIRI/bevacizumab
Drug: Placebo — Dextrose 5% in water or normal saline (sodium chloride solution 0.9%) administered by IV infusion over 30 (±10) minutes no more than 4 hours prior to each Day 1 chemotherapy administration. Second dose of placebo was administered on Day 2.
  Arms: placebo + FOLFOXIRI/bevacizumab

SUMMARY:
This was a randomized, double-blind, placebo-controlled, global, multicenter, Phase 3 trial evaluating the impact of trilaciclib on myelopreservation and anti-tumor efficacy when administered prior to FOLFOXIRI/bevacizumab in patients with pMMR/MSS mCRC who have not received systemic therapy for metastatic disease.

DETAILED DESCRIPTION:
Patients were randomly assigned (1:1) to receive placebo or trilaciclib on Days 1 and 2 administered intravenously (IV) prior to FOLFOXIRI/bevacizumab in 14-day cycles for up to 12 cycles (Induction).

Following completion of Induction, patients continued in Maintenance, where they received trilaciclib or placebo per randomization allocation at study entry. Trilaciclib/placebo will be administered prior to infusional-5FU/leucovorin/bevacizumab at the same dose and schedule used during Induction. The patient continued to receive treatment on study until disease progression, unacceptable toxicity, withdrawal of consent, discontinuation by Investigator, or the end of the trial, whichever occurs first. Treatment cycles occurred consecutively without interruption, except when necessary to manage toxicities or for administrative reasons.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years of age at the time of signing the informed consent. Patients > 70 years of age must have a G8 Health State Screening Tool (geriatric screening tool) score > 14.
2. Proficient mismatch repair/microsatellite stable (pMMR/MSS), histologically or cytologically-confirmed adenocarcinoma of the colon or rectum. Patients with any BRAF or KRAS mutation status (wild type or mutant) are eligible. If historical pMMR/MSS and/or BRAF V600E mutational status are not known, a tumor specimen (archival or fresh biopsy) must be sent for testing and results must be available at the time of randomization in interactive web response system (IWRS). If testing cannot be completed using a standard clinical assay performed institutionally/locally, the tumor specimen may be sent to the Sponsor's designated central laboratory for analysis; only historical KRAS mutational status will be collected (ie, no testing required prior to study entry). Note: Any sample sent for MSS/BRAF analysis will be in addition to that required per Inclusion Criterion 5.
3. Unresectable and measurable or metastatic colorectal cancer per RECIST v1.1
4. ECOG performance status of 0 to 1
5. A formalin-fixed paraffin-embedded (FFPE) tumor specimen (from archival or fresh biopsy) with an associated pathology report documenting pMMR/MSS mCRC must be confirmed to be available to send to the Sponsor for planned retrospective biomarker analyses (tissue requirements are provided in the associated laboratory manual).
6. Hemoglobin ≥ 9.0 g/dL in the absence of RBC transfusion or ESA administration within 14 days prior to first dose of trilaciclib/placebo
7. Absolute neutrophil count (ANC) ≥ 1.5 × 10^9 /L
8. Platelet count ≥ 100 × 10^9 /L
9. Estimated glomerular filtration rate (eGFR) ≥ 30 mL/minute/1.73m^2
10. Total bilirubin ≤ 1.5 × upper limit of normal (ULN)
11. AST, ALT, and alkaline phosphatase ≤ 3 × ULN for patients without liver or bone metastases; AST, ALT and alkaline phosphatase ≤ 5 × ULN in the presence of liver metastases; AST and ALT ≤ 3 x ULN and alkaline phosphatase ≤ 5 × ULN in the presence of bone metastases
12. Resolution of nonhematologic toxicities from prior therapy or surgical procedures to ≤ Grade 1 or baseline (except alopecia)
13. Urine dipstick protein < 2+. If ≥ 2+ at Screening, then a 24-hour urine collection must be done to demonstrate ≤ 1 g of protein/24 hours
14. Contraceptive use by men or women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies. Please see Section 17.4 for detailed instructions on methods of contraception requirements.
15. Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.

Exclusion Criteria:

1. Prior systemic therapy for mCRC. Patients who received adjuvant/neoadjuvant therapy (ie, treatment with curative intent) for colorectal cancer are eligible if it has been ≥ 6 months between the last dose of systemic chemotherapy and the date of informed consent.
2. Any radiotherapy, chemotherapy, immunotherapy, biologic, investigational, or hormonal therapy for cancer treatment (except for adjuvant hormonal therapy for breast cancer or prostate cancer defined as M0 disease or PSA persistence/recurrence without metastatic disease) within 3 weeks prior to the first dose of trilaciclib/placebo.
3. Receipt of any low-dose systemic chemotherapeutic agent (e.g., low-dose methotrexate for rheumatoid arthritis) administered for a nononcologic purpose within 3 weeks prior to the first dose of trilaciclib/placebo.
4. Presence of central nervous system (CNS) metastases/leptomeningeal disease requiring immediate treatment with radiation therapy or steroids (i.e., patient must be off steroids administered for brain metastases for at least 14 days prior to the first dose of trilaciclib/placebo).
5. QTcF interval > 450 msec (males) or > 470 msec (females) at screening. For patients with ventricular pacemakers, QTcF > 500 msec.
6. Personal or family history of long QT syndrome
7. Symptomatic peripheral neuropathy
8. History of interstitial lung disease (ILD)
9. Uncontrolled hypertension (blood pressure ≥ 150/90mm Hg)
10. Clinically significant (i.e., active) cardiovascular disease at the time of signing the informed consent; for example cerebrovascular accidents (≤ 6 months before the first dose of trilaciclib/placebo), myocardial infarction (≤ 6 months before the first dose of trilaciclib/placebo), unstable angina, serious cardiac arrhythmia requiring medication, or uncontrolled symptomatic congestive heart failure [Class II or higher as defined by the New York Heart Association [NYHA] functional classification system])
11. Serious, non-healing wound, ulcer, or bone fracture
12. Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to study treatment start, or anticipation of the need for major surgical procedure during the course of the study.
13. Known serious active infection (e.g., human immunodeficiency virus [HIV], hepatitis B or C, tuberculosis, etc.)
14. Known Gilbert's Syndrome or homozygous for the UGT1A1*28 allele. UGT1A1 genotyping is not required for this study.
15. Chronic inflammatory bowel disease and/or active intestinal obstruction. Patients should not be treated until the intestinal obstruction has resolved.
16. Previous history of significant/severe hemorrhage, within 1 month before randomization. History of previous abdominal fistula or gastrointestinal perforation within 6 months before randomization
17. Known history of bleeding diathesis or coagulopathy
18. INR > 1.5 within 14 days prior to starting study treatment. EXEMPTION: patients on full anticoagulation must have an in-range INR (usually between 2 to 3) if INR is used for monitoring. Any anticoagulation therapy must be at stable dosing prior to enrollment.
19. Ongoing or anticipated treatment with potent cytochrome inhibitors CYP450 3A4 (such as ketoconazole) or inducers (such as rifampicin, carbamazepine, phenobarbital, phenytoin or St. John's wort). Irinotecan should not be delivered concurrently.
20. Patients with ongoing or anticipated treatment with sorivudine or its chemically related analogues, such as brivudine.
21. Chronic, daily treatment with high-dose aspirin (> 325 mg/day)
22. Prior allogeneic or autologous hematopoietic stem cell or bone marrow transplantation
23. Receipt of any live attenuated vaccines within 4 weeks prior to first dose of study treatment
24. Known hypersensitivity to any of the drugs used in this study
25. Pregnant or lactating women
26. Legal incapacity or limited legal capacity
27. Other uncontrolled serious chronic disease or psychiatric condition that in the Investigator's opinion could affect patient safety, compliance, or follow-up in the protocol
28. Any contraindications to the administration of FOLFOXIRI and bevacizumab at the discretion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 326 (Actual)
Dates: Start 2021-01-06 (Actual); Primary Completion 2023-02-13 (Actual); Study Completion 2023-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Contact, Study Director — G1 Therapeutics, Inc.
Locations (82):
- United States (24):
  - AZ Oncology Associates - HOPE, Tucson, Arizona
  - Beverly Hills Cancer Center, Beverly Hills, California
  - Keck Medical Center of USC Pasadena, Los Angeles, California
  - The Oncology Institute of Hope & Innovation\ Innovative Clinical Research Institute, Whittier, California
  - Georgetown University - Lombardi Comprehensive Cancer Center, Washington D.C., District of Columbia
  - Florida Cancer Specialists (South Region), Fort Myers, Florida
  - Florida Cancer Specialists NORTH, Fort Myers, Florida
  - Mid-Florida Hematology & Oncology Centers, P.A., Orange City, Florida
  - Florida Cancer Specialists, St. Petersburg, Florida
  - Florida Cancer Specialists - Panhandle, Tallahassee, Florida
  - Northside Hospital - Georgia Cancer Specialists, Atlanta, Georgia
  - Illinois Cancer Specialists, Arlington Heights, Illinois
  - Boston Medical Center, Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Comp. Cancer Centers of Nevada, Las Vegas, Nevada
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oregon Health & Science University, Portland, Oregon
  - Gettysburg Cancer Center, Gettysburg, Pennsylvania
  - Tennessee Oncology, Nashville, Tennessee
  - UT Southwestern Medical Center, Dallas, Texas
  - Millennium Oncology, Kingswood, Texas
  - Inova Schar Cancer Institute, Fairfax, Virginia
  - Onc and Hem Assoc of SW VA, Roanoke, Virginia
- China (10):
  - Henan Cancer Hospital, Zijingshan, Henan
  - Wuhan Union Hospital, Wuhan, Hubei
  - Jilin Provincial Tumor Hospital, Changchun, Jilin
  - The First Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - The Affiliated Tumor Hospital of Harbin Medical University, Heilongjiang
  - Jinan Central hospital, Shandong
  - Zhongshan Hospital Fudan University, Shanghai
  - Xuzhou Central hospital, Xuzhou
  - First Affiliated Hospital of Zhengzhou University, Zhengzhou
- Hungary (4):
  - Orszagos Onkologiai Intezet, Budapest
  - Bekes Megyei Kozponti Korhaz Pandy Kalman Tagkorhaza, Gyula
  - Bacs-Kiskun Megyei Oktatokorhaz, Kecskemét
  - SzSzB Megyei Korhazak es Egyetemi Oktatokorhaz, Nyíregyháza
- Italy (5):
  - ASL Regionale Piemonte - Ospedale Santo Spirito Casale Monferrato (Ospedale di Casale Monferrato), Casale Monferrato, Alessandria
  - Azienda Ospedaliera Universitaria Policlinico Tor Vergata, Rome, Roma
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome, Roma
  - Fondazione IRCCS CA' Granda Ospedale Maggiore Policlinico, Cremona
  - Azienda Ospedaliera Universitaria Careggi, Florence
- Poland (5):
  - Szpitale Pomorskie spółka z ograniczoną odpowiedzialnością, Gdynia
  - Szpital Specjalistyczny im. L.Rydygiera w Krakowie, Krakow
  - Mrukmed Lekarz Beata Madej Mruk i Partner Spółka Partnerska Oddział nr 1 w Rzeszowie, Rzeszów
  - Centrum Medyczne Pratia Poznan, Skórzewo
  - Centrum Zdrowia MDM, Warsaw
- Spain (15):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - ICO l'Hospitalet - Hospital Duran i Reynals, Barcelona
  - Hospital Universitari Arnau de Vilanova, Lleida
  - Hospital Universitario Lucus Augsti, Lugo
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario HM Madrid Sanchinarro, Madrid
  - Hospital Universitario Puerta de Hierro Majadahonda, Madrid
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Clinico Universitario de Valencia, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza
- Ukraine (15):
  - CI Cherkasy Regional Oncological Dispensary of CRC, Cherkasy
  - MI Regional Clinical Oncologycal Dispensary, Dnipro
  - Dnipropetrovsk City Multispecialty Clinical Hospital #4, Dnipro
  - Limited Liability Company "Medical Center named by Academician Yuriy Prokopovich Spizhenko", Kapitanivka
  - CNE Prof. O.O. Shalimov Kharkiv City Clinical Hospital #2 of KCC, Kharkiv
  - Communal Non-profit Enterprise Regional Center of Oncology, Kharkiv NMU, Kharkiv
  - Treatment-Diagnostic Center of Private Enterprise of PPC Atsynus, Kropyvnytskyi
  - CI Kryvyi Rih Oncological Dispensary of DRC, Kryvyi Rih
  - Medical Center Asklepion LLC, Kyiv
  - Medical Center of Limited Liability Company Medical Center Concilium Medical, Kyiv
  - Communal Enterprise Volyn Regional Medical Center of Oncology of Volyn Regional Council, Lutsk
  - Communal Institution Odesa Regional Clinical Hospital; Department of Surgery, Odesa
  - University Hospital of Sumy State University, Sumy
  - CNE CCCH of Uzh CC Oncological Center, Ther Dept, SHEI UNU, Uzhhorod
  - Medical center "Oncolife" LLC, Zaporizhzhia
- United Kingdom (4):
  - Barts Hospital, London, Greater London
  - Royal Free Hospital, London, Greater London
  - The Christie, Manchester, Greater Manchester
  - Velindre Cancer Centre, Cardiff, South Glamorgan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lenz HJ, Liu T, Chen EY, Horvath Z, Bondarenko I, Danielewicz I, Ghidini M, Garcia-Alfonso P, Jones R, Aapro M, Zhang Y, Wang J, Wang W, Adeleye J, Beelen A, Hubbard J. Trilaciclib prior to FOLFOXIRI/bevacizumab for patients with untreated metastatic colorectal cancer: phase 3 PRESERVE 1 trial. JNCI Cancer Spectr. 2025 Jan 3;9(1):pkae116. doi: 10.1093/jncics/pkae116. PMID 39579142

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 89 study centers in 8 countries consented at least 1 participant. The first participant was enrolled on January 6, 2021 and the last visit of the last participant occurred on March 31, 2023.
Pre-assignment Details: A total of 458 participants were screened in this study. 326 participants were randomized in a double-blind manner to receive either trilaciclib or placebo, administered on Days 1 and 2 of each cycle of FOLFOXIRI and bevacizumab therapy. A total of 319 participants received at least 1 dose of study drug.
Groups:
- Trilaciclib + FOLFOXIRI/Bevacizumab: During Induction the following study drugs were administered on Day 1:
  Trilaciclib - IV infusion prior to chemotherapy Irinotecan- IV, Oxaliplatin - IV, Leucovorin- IV, Fluorouracil (5-FU) - continuous infusion (CI) over 46-48 hours beginning on Day 1, Bevacizumab - IV
  The Induction Day 1 administration of trilaciclib was repeated on Induction Day 2.
  Following completion of Induction, patients continued in Maintenance, where they continued to receive trilaciclib per randomization allocation. Trilaciclib was administered prior to infusional-5FU/leucovorin/bevacizumab at the same dose and schedule used during Induction.
- Placebo + FOLFOXIRI/Bevacizumab: The subjects in the placebo arm followed the same schedule as the trilaciclib arm, but received placebo instead of trilaciclib
  Placebo: dextrose 5% in water or normal saline (sodium chloride solution 0.9%)
Period: Overall Study
Arm/Group | Trilaciclib + FOLFOXIRI/Bevacizumab | Placebo + FOLFOXIRI/Bevacizumab
Started (All patients in the ITT population.) | 164 | 162
Patients With ≥ 1 Dose of Study Drug, n (%) | 159 | 160
Completed | 0 | 0
Not Completed | 164 | 162
Not completed — Death | 49 | 26
Not completed — Lost to Follow-up | 3 | 4
Not completed — Study terminated by Sponsor | 92 | 114
Not completed — Withdrawal by Subject | 12 | 11
Not completed — Other, unspecified | 8 | 7

BASELINE CHARACTERISTICS:
Population: Information presented is based on overall enrollment into the study and constitutes the ITT population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Trilaciclib + FOLFOXIRI/Bevacizumab | Placebo + FOLFOXIRI/Bevacizumab | Total
Number analyzed (Participants) | 164 | 162 | 326
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.2 (11.80) | 55.5 (10.60) | 55.8 (11.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 61 | 119
  Male | 106 | 101 | 207
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 119 | 112 | 231
  Black or African American | 4 | 9 | 13
  Asian | 32 | 33 | 65
  Other | 3 | 0 | 3
  Not Reported | 3 | 3 | 6
  Unknown | 3 | 5 | 8

OUTCOME MEASURES:

1. Primary Outcome: Duration of Severe Neutropenia (DSN)
Description: The DSN was defined as the number of days for the first severe neutropenia (SN) event in Cycles 1, 2, 3, or 4 for participants who had at least one SN event in the first 4 cycles of Induction. It was calculated as the days from the date of the first absolute neutrophil count (ANC) value of < 0.5 × 10^9/L to the date of the first ANC value ≥ 0.5 × 10^9/L where no additional ANC values < 0.5 × 10^9/L were observed for the remainder of that cycle.
Time Frame: Cycles 1 to 4 (14-day cycles up to 56 days)
Population: A Modified Intent-to-Treat (mITT) population was utilized in order to account for potential data integrity issues resulting from the war in Ukraine. The criteria for patients to be included in the mITT population consisted of all patients being randomized in countries other than Ukraine and all patients in Ukraine being randomized prior to 09 September 2021.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Trilaciclib + FOLFOXIRI/Bevacizumab | Placebo + FOLFOXIRI/Bevacizumab
Number analyzed (Participants) | 149 | 147
days | 0.1 (0.84) | 1.3 (3.14)
Statistical Analysis 1: Comparison: Trilaciclib + FOLFOXIRI/Bevacizumab vs Placebo + FOLFOXIRI/Bevacizumab; Test type: Other; p < 0.001, ANCOVA — Two-sided p-value for treatment effect was generated from a nonparametric ANCOVA controlling for stratification factors of Region and Prior chemotherapy with study baseline ANC value as a covariate; Mean Difference (Final Values) = -1.2, 95% CI 2-sided [-1.7 to -0.6]

2. Primary Outcome: Occurrence of Severe Neutropenia (SN) During Induction
Description: Severe neutropenia was defined as the absolute neutrophil count (ANC) laboratory value that met the Common Terminology Criteria for Adverse vents (CTCAE) criteria for ≥ Grade 4 toxicity (ie, ANC < 0.5 × 10^9/L in SI Unit)
Time Frame: Induction Period, cycles 1-12 (14-day cycles up to 168 days)
Population: as for outcome 1
Measure: Number; unit: event per 100 cycles
Arm/Group | Trilaciclib + FOLFOXIRI/Bevacizumab | Placebo + FOLFOXIRI/Bevacizumab
Number analyzed (Participants) | 149 | 147
event per 100 cycles | 0.1 | 3
Statistical Analysis 1: Comparison: Trilaciclib + FOLFOXIRI/Bevacizumab; Test type: Other; p < 0.001, modified Poisson model; aRR = 0.04, 95% CI 2-sided [0.01 to 0.19], Standard Error of Mean 0.032

3. Secondary Outcome: Overall Survival (OS)
Description: Overall survival is defined as the time from the date of the first dose of study treatment to the date of death from any cause.
Time Frame: Up to 52 months
Population: Due to early study termination, data were not collected for this outcome measure.
Arm/Group | Trilaciclib + FOLFOXIRI/Bevacizumab | Placebo + FOLFOXIRI/Bevacizumab
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Additional Myelopreservation Measures
Description: To assess the effects of trilaciclib on additional measures of the neutrophil lineage compared with placebo in patients receiving FOLFOXIRI/bevacizumab for pMMR/MSS mCRC as measured by the number of SN events, granulocyte-colony stimulating factor (G-CSF) administration and febrile neutropenia (FN) adverse events (AE)
Time Frame: Through Induction Period - on average 24 weeks (up to 12 cycles) of FOLFOXIRI/bevacizumab
Population: Due to early study termination, data were not collected for this outcome measure.
Arm/Group | Trilaciclib + FOLFOXIRI/Bevacizumab | Placebo + FOLFOXIRI/Bevacizumab
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Red Blood Cell Lineage
Description: To assess the effects of trilaciclib on the red blood cell (RBC) lineage compared with placebo in patients receiving FOLFOXIRI/bevacizumab for pMMR/MSS mCRC by measure of Grade 3 or 4 decreased hemoglobin laboratory values, RBC transfusions on or after Week 5, and erythropoiesis-stimulating agents (ESA) administration
Time Frame: Through Induction Period - on average 24 weeks (up to 12 cycles) of FOLFOXIRI/bevacizumab
Population: Due to early study termination, data were not collected for this outcome measure.
Arm/Group | Trilaciclib + FOLFOXIRI/Bevacizumab | Placebo + FOLFOXIRI/Bevacizumab
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Platelet Lineage
Description: To assess the effects of trilaciclib on the platelet lineage compared with placebo in patients receiving FOLFOXIRI/bevacizumab for pMMR/MSS mCR by measure of Grade 3 or 4 decreased platelet count laboratory values and Platelet transfusions.
Time Frame: Through Induction Period - on average 24 weeks (up to 12 cycles) of FOLFOXIRI/bevacizumab
Population: Due to early study termination, data were not collected for this outcome measure.
Arm/Group | Trilaciclib + FOLFOXIRI/Bevacizumab | Placebo + FOLFOXIRI/Bevacizumab
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Multiple Lineage
Description: To assess the effects of trilaciclib on multiple lineages compared with placebo in patients receiving FOLFOXIRI/bevacizumab for pMMR/MSS mCRC by measure of Grade 3 or 4 hematologic lab values.
Time Frame: Through Induction Period - on average 24 weeks (up to 12 cycles) of FOLFOXIRI/bevacizumab
Population: Due to early study termination, data were not collected for this outcome measure.
Arm/Group | Trilaciclib + FOLFOXIRI/Bevacizumab | Placebo + FOLFOXIRI/Bevacizumab
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Standard of Care Dosing
Description: To assess the effects of trilaciclib on standard of care dosing compared with placebo in patients receiving FOLFOXIRI/ bevacizumab for pMMR/MSS mCRC by measure of all-cause dose reductions or cycle delays and relative dose intensity for FOLFOXIRI/bevacizumab
Time Frame: Through Induction Period - on average 24 weeks (up to 12 cycles) of FOLFOXIRI/bevacizumab
Population: Due to early study termination, data were not collected for this outcome measure.
Arm/Group | Trilaciclib + FOLFOXIRI/Bevacizumab | Placebo + FOLFOXIRI/Bevacizumab
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Healthcare Utilization
Description: To assess the effects of trilaciclib on healthcare utilization compared with placebo in patients receiving FOLFOXIRI/ bevacizumab for pMMR/MSS mCRC by measure of hospitalizations and antibiotic use.
Time Frame: Through Induction Period - on average 24 weeks (up to 12 cycles) of FOLFOXIRI/bevacizumab
Population: Due to early study termination, data were not collected for this outcome measure.
Arm/Group | Trilaciclib + FOLFOXIRI/Bevacizumab | Placebo + FOLFOXIRI/Bevacizumab
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Best Overall Response (BOR)
Description: Best overall response (BOR) will be determined using all visit responses prior to or on the date of (i) radiographic disease progression; (ii) withdrawal of consent to obtain scans; (iii) death; (iv) lost to follow-up; or (v) initiation of subsequent anti-cancer therapy other than the study drugs, whichever is earlier will be based on RECIST v1.1.
Time Frame: Through Induction Period - on average 24 weeks (up to 12 cycles) of FOLFOXIRI/bevacizumab
Population: The Response Evaluable (RE) population included those patients in the mITT population who received at least 1 dose of any study drug and had measurable (target) tumor lesion(s) at the baseline tumor assessment. The patients also had at least 1 post-baseline tumor assessment, discontinued treatment because of clinical progression prior to their first post-baseline tumor scan, or died due to disease progression prior to their first post-baseline tumor scan.
Measure: Number; unit: percentage of participants
Arm/Group | Trilaciclib + FOLFOXIRI/Bevacizumab | Placebo + FOLFOXIRI/Bevacizumab
Number analyzed (Participants) | 137 | 140
percentage of participants
  Complete response | 0 | 3
  Partial response | 75 | 91
  Stable disease | 50 | 36
  Progressive disease | 5 | 7
  Not evaluable | 7 | 3

11. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR was defined as the percentage of participants in the analysis population who had a Complete Response (CR) defined as a disappearance of all target lesions with pathological lymph nodes having a reduction in short axis to <10 mm or Partial Response (PR) defined as at least a 30% decrease in the sum of diameters of target lesions, using the baseline sum diameters as a reference based on RECIST v1.1.
Time Frame: Assessed from the day of the first dose of the study drug, through 30 days after the last dose of the study drug, up to 115 weeks
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Trilaciclib + FOLFOXIRI/Bevacizumab | Placebo + FOLFOXIRI/Bevacizumab
Number analyzed (Participants) | 137 | 140
percentage of participants | 41.6 [33.3 to 50.3] | 57.1 [48.5 to 65.5]

12. Secondary Outcome: Duration of Objective Response (DOR)
Description: DOR is the time between first objective response of CR or PR and the first date that progressive disease is objectively documented or death, whichever comes first.
Time Frame: as for outcome 11
Population: as for outcome 10
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Trilaciclib + FOLFOXIRI/Bevacizumab | Placebo + FOLFOXIRI/Bevacizumab
Number analyzed (Participants) | 137 | 140
months | 9.1 [7.9 to 10.2] | 12.7 [9.5 to NA] — The upper limit of the 95% Confidence Interval was not estimable due to insufficient participants with events.

13. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the time from the date of randomization until the date of documented radiologic disease progression per RECIST v1.1 or death due to any cause, whichever comes first.
Time Frame: as for outcome 11
Population: Modified Intent-to-Treat (mITT) population was utilized in order to account for potential data integrity issues resulting from the war in Ukraine. The criteria for patients to be included in the mITT population consisted of all patients being randomized in countries other than Ukraine and all patients in Ukraine being randomized prior to 09 September 2021.
Measure: Mean (95% Confidence Interval); unit: months
Arm/Group | Trilaciclib + FOLFOXIRI/Bevacizumab | Placebo + FOLFOXIRI/Bevacizumab
Number analyzed (Participants) | 149 | 147
months | 10.3 [8.6 to 11] | 13.1 [11 to 18.5]

14. Secondary Outcome: Quality of Life/ Effects on Chemotherapy-Induced Fatigue
Description: To assess the effects of trilaciclib on chemotherapy-induced fatigue compared with placebo in patients receiving FOLFOXIRI/bevacizumab for pMMR/MSS mCRC, as measured by Time To First Confirmed Deterioration of Fatigue (TTCD-fatigue) during Induction, as measured by the FACIT-F (Functional Assessment of Chronic Illness Therapy-Fatigue).
Time Frame: Through Induction Period- on average 24 weeks (up to 12 cycles) of FOLFOXIRI/bevacizumab
Population: Due to early study termination, data were not collected for this outcome measure.
Arm/Group | Trilaciclib + FOLFOXIRI/Bevacizumab | Placebo + FOLFOXIRI/Bevacizumab
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Number of Participants With Reported Adverse Events to Measure Safety and Tolerability
Description: To assess the safety and tolerability of trilaciclib compared with placebo in patients receiving FOLFOXIRI/ bevacizumab for pMMR/MSS mCRC by measure of occurrence and severity of AEs by National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) v5.0, changes in laboratory parameters, vital signs and electrocardiogram (ECG) parameters, grade 3 or 4 abnormalities in chemistry laboratory parameters, and study treatment discontinuation due to AEs.
Time Frame: Safety was assessed from the day of the first dose of the study drug, through 30 days after the last dose of the study drug, up to 115 weeks
Population: The Safety population included all randomized patients who received at least 1 dose of any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Trilaciclib + FOLFOXIRI/Bevacizumab | Placebo + FOLFOXIRI/Bevacizumab
Number analyzed (Participants) | 159 | 160
Participants
  Number of patients with any AE | 157 | 159
  Number of patients with any AE of CTCAE Grade ≥ 3 | 106 | 117
  Number of patients with any AE of CTCAE Grade ≥ 4 | 18 | 35
  Number of patients with any study drug-related AE | 154 | 155
  Trilaciclib/Placebo-Related AE | 109 | 103
  Fluorouracil-related AE | 139 | 151
  Leucovorin-related AE | 103 | 122
  Oxaliplatin-related AE | 143 | 151
  Irinotecan-related AE | 143 | 151
  Bevacizumab-related AE | 127 | 128
  Patients with any serious AE | 47 | 47
  Patients with AE leading to discontinuation of any study drug | 50 | 47
  Leading to trilaciclib/placebo discontinuation | 19 | 13
  Leading to fluorouracil discontinuation | 19 | 14
  Leading to leucovorin discontinuation | 20 | 13
  Leading to oxaliplatin discontinuation | 38 | 30
  Leading to irinotecan discontinuation | 20 | 20
  Leading to bevacizumab discontinuation | 31 | 26
  Patients with trilaciclib/placebo-related AE leading to discontinuation of any study drug | 10 | 9
  Patients with AE leading to death | 8 | 3
  Patients with AESI for trilaciclib | 33 | 28

ADVERSE EVENTS:
Time Frame: Safety was assessed from the day of the first dose of the study drug, through 30 days after the last dose of the study drug, up to 115 weeks.
Description: Analysis was performed on the Safety analysis set which included all randomized participants who received at least one dose of any study drug.
Arm/Group | Trilaciclib + FOLFOXIRI/Bevacizumab | Placebo + FOLFOXIRI/Bevacizumab
All-Cause Mortality (participants affected / at risk) | 49/159 | 26/160
Serious Adverse Events (participants affected / at risk) | 47/159 | 47/160
Other Adverse Events (participants affected / at risk) | 155/159 | 159/160
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Trilaciclib + FOLFOXIRI/Bevacizumab (N=159) | Placebo + FOLFOXIRI/Bevacizumab (N=160)
Anaemia (Blood and lymphatic system disorders) | 0 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 5
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 5
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Cardiac failure acute (Cardiac disorders) | 1 | 0
Left ventricular dysfunction (Cardiac disorders) | 0 | 1
Myocardial injury (Cardiac disorders) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 1
Abdominal adhesions (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 3
Anal fistula (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 3
Enterocutaneous fistula (Gastrointestinal disorders) | 1 | 0
Gastrointestinal obstruction (Gastrointestinal disorders) | 1 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 2 | 1
Ileus paralytic (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 4 | 3
Intestinal perforation (Gastrointestinal disorders) | 1 | 1
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 0 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 1
Oesophageal rupture (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 2 | 0
Rectal perforation (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Subileus (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 3 | 2
Death (General disorders) | 1 | 0
Device related thrombosis (General disorders) | 1 | 0
Pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 3
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Drug hypersensitivity (Immune system disorders) | 1 | 0
Abdominal abscess (Infections and infestations) | 1 | 0
Abscess limb (Infections and infestations) | 0 | 1
Anal abscess (Infections and infestations) | 0 | 1
Anorectal infection (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 0 | 1
COVID-19 (Infections and infestations) | 1 | 1
COVID-19 pneumonia (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 2
Device related infection (Infections and infestations) | 0 | 1
Infectious pleural effusion (Infections and infestations) | 1 | 0
Intestinal sepsis (Infections and infestations) | 1 | 0
Neutropenic sepsis (Infections and infestations) | 0 | 1
Pelvic abscess (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 3 | 1
Pyelonephritis (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 3
Drain site complication (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 1
Blood bilirubin increased (Investigations) | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Myopathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0
Lumbar radiculopathy (Nervous system disorders) | 1 | 0
Myoclonic epilepsy (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 1
Anxiety (Psychiatric disorders) | 0 | 1
Completed suicide (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Pulmonary thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Aortic embolus (Vascular disorders) | 1 | 0
Embolism (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 1
Jugular vein thrombosis (Vascular disorders) | 0 | 1
Superior vena cava syndrome (Vascular disorders) | 0 | 1
Thrombosis (Vascular disorders) | 0 | 1
Venous thrombosis (Vascular disorders) | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Trilaciclib + FOLFOXIRI/Bevacizumab (N=159) | Placebo + FOLFOXIRI/Bevacizumab (N=160)
Anaemia (Blood and lymphatic system disorders) | 57 | 61
Leukopenia (Blood and lymphatic system disorders) | 27 | 35
Neutropenia (Blood and lymphatic system disorders) | 61 | 92
Thrombocytopenia (Blood and lymphatic system disorders) | 34 | 36
Abdominal distension (Gastrointestinal disorders) | 9 | 6
Abdominal pain (Gastrointestinal disorders) | 34 | 36
Abdominal pain upper (Gastrointestinal disorders) | 9 | 8
Constipation (Gastrointestinal disorders) | 38 | 29
Diarrhoea (Gastrointestinal disorders) | 83 | 118
Dyspepsia (Gastrointestinal disorders) | 11 | 10
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 10 | 6
Haemorrhoids (Gastrointestinal disorders) | 5 | 11
Nausea (Gastrointestinal disorders) | 85 | 101
Oral dysaesthesia (Gastrointestinal disorders) | 5 | 8
Rectal haemorrhage (Gastrointestinal disorders) | 7 | 9
Stomatitis (Gastrointestinal disorders) | 25 | 42
Vomiting (Gastrointestinal disorders) | 54 | 64
Asthenia (General disorders) | 28 | 28
Fatigue (General disorders) | 53 | 52
Mucosal inflammation (General disorders) | 17 | 18
Pyrexia (General disorders) | 17 | 22
Temperature intolerance (General disorders) | 10 | 5
COVID-19 (Infections and infestations) | 18 | 22
Upper respiratory tract infection (Infections and infestations) | 7 | 12
Urinary tract infection (Infections and infestations) | 11 | 10
Alanine aminotransferase increased (Investigations) | 20 | 24
Aspartate aminotransferase increased (Investigations) | 20 | 24
Blood alkaline phosphatase increased (Investigations) | 13 | 11
Gamma-glutamyltransferase increased (Investigations) | 9 | 9
Neutrophil count decreased (Investigations) | 12 | 15
Platelet count decreased (Investigations) | 9 | 7
Weight decreased (Investigations) | 20 | 29
White blood cell count decreased (Investigations) | 8 | 12
Decreased appetite (Metabolism and nutrition disorders) | 36 | 39
Dehydration (Metabolism and nutrition disorders) | 12 | 11
Hyperglycaemia (Metabolism and nutrition disorders) | 11 | 8
Hypoalbuminaemia (Metabolism and nutrition disorders) | 6 | 11
Hypokalaemia (Metabolism and nutrition disorders) | 21 | 21
Hypomagnesaemia (Metabolism and nutrition disorders) | 9 | 3
Hypophosphataemia (Metabolism and nutrition disorders) | 6 | 12
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 13
Back pain (Musculoskeletal and connective tissue disorders) | 9 | 11
Muscle spasms (Musculoskeletal and connective tissue disorders) | 20 | 9
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 | 6
Dizziness (Nervous system disorders) | 13 | 19
Dysgeusia (Nervous system disorders) | 12 | 10
Headache (Nervous system disorders) | 32 | 26
Neuropathy peripheral (Nervous system disorders) | 36 | 26
Neurotoxicity (Nervous system disorders) | 10 | 13
Paraesthesia (Nervous system disorders) | 20 | 15
Peripheral sensory neuropathy (Nervous system disorders) | 37 | 34
Tremor (Nervous system disorders) | 8 | 1
Anxiety (Psychiatric disorders) | 13 | 12
Insomnia (Psychiatric disorders) | 15 | 15
Proteinuria (Renal and urinary disorders) | 19 | 25
Cough (Respiratory, thoracic and mediastinal disorders) | 13 | 12
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11 | 8
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 7 | 28
Hiccups (Respiratory, thoracic and mediastinal disorders) | 14 | 9
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 10 | 6
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 | 8
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4 | 10
Alopecia (Skin and subcutaneous tissue disorders) | 23 | 25
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 4 | 8
Hypertension (Vascular disorders) | 34 | 35
Hypotension (Vascular disorders) | 5 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator will submit results communications for review by the sponsor at least 60 days prior to expected submission to the intended publisher or meeting committee. This review period may be shortened upon mutual consent. The sponsor may request modification of any publication, presentation or use by the investigator if such activity may jeopardize a patent application, an existing patent, or other proprietary rights.

DOCUMENTS (2):
  • Study Protocol (2022-12-15): https://cdn.clinicaltrials.gov/large-docs/68/NCT04607668/Prot_000.pdf
  • Statistical Analysis Plan (2023-01-09): https://cdn.clinicaltrials.gov/large-docs/68/NCT04607668/SAP_001.pdf